CLINICAL TRIAL: NCT02148419
Title: Psychosocial Development of Maltreated Children: A Prospective Study
Status: Terminated | Type: Observational
Why Stopped: recruiting not successful, too few participants
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Andreas Jud,PhD, Dr. Andreas Jud, University Children's Hospital, Zurich
Other Study IDs: KEK-ZH-Nr. 2013-0331
Record Dates: First submitted 2014-05-13; First posted 2014-05-28 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Quality of Life
Keywords: quality of life; maltreatment; neglect; childhood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
Between 2007-2010 the Child Protection Team (CPT) at University Children's Hospital Zurich was the first in Europe to follow up the development of maltreated children in a hospital sample . The follow-up took place 2-3 years after the child had been reported to the CPT. As a major result, children's health-related quality of life (HRQoL) had been impaired in maltreated children compared to controls (Jud, Landolt, Tatalias, Lach, & Lips, 2012). However, this difference only emerged for the self-assessment of HRQoL by children aged 6 years or older .To address limitations, the CPT at University Children's Hospital Zurich and Children's Hospital Baden AG propose a prospective study with a baseline at the time of report to the CPT and a two year follow-up. This study aims at analyzing HRQoL, behavior and mental health of maltreated children prospectively and will be the first to provide data on changes in HRQoL in the aftermath of maltreatment. We assume the following hypotheses:

* The HRQoL and mental health of children will be impaired following maltreatment even while controlling for others possible predictors of impaired HRQoL and mental health.
* We assume a dose-response relationship between severity of maltreatment and impaired HRQoL. Multiple maltreatment is hypothesized to have a larger impact then a single type of maltreatment.
* At baseline, HRQoL scores are hypothesized to be at a markedly low level. We assume a slight increase in HRQoL from baseline to first follow-up, but not a continuing increase to second follow-up.

DETAILED DESCRIPTION:
Between 2007-2010 the Child Protection Team (CPT) at University Children's Hospital Zurich was the first in Europe to follow up the development of maltreated children in a hospital sample (Jud, Lips, & Landolt, 2010). Out of a total 180 children in the 2005/2006 CPT caseload, 42 children between 2.5 and 16.5 years and their primary caregiver participated (Jud, Lips, et al., 2010). The follow-up took place 2-3 years after the child had been reported to the CPT. Non-CPT reported hospital patients were used as controls, matched for age, gender, nationality, and medical condition. As a major result, children's health-related quality of life (HRQoL) had been impaired in maltreated children compared to controls (Jud, Landolt, Tatalias, Lach, & Lips, 2012). However, this difference only emerged for the self-assessment of HRQoL by children aged 6 years or older (Jud et al., 2012). The assessment of children's HRQoL by primary caregivers showed no significant differences for maltreated children compared to controls for all age groups. An essential lack of understanding of the child's experiences and beliefs is not only likely to affect the child's HRQoL, but may also contribute to cur-rent and future risk of maltreatment (Jud et al., 2012). Furthermore, maltreated children had increased depression scores and more behavior problems compared to controls. Detailed results can be found in Jud et al. (Jud et al., 2012; Jud, Lips, et al., 2010). To address these limitations, the CPT at University Children's Hospital Zurich and Children's Hospital Baden AG propose a prospective study with a baseline at the time of report to the CPT and a two year follow-up. This study aims at analyzing HRQoL, behavior and mental health of maltreated children prospectively and will be the first to provide data on changes in HRQoL in the aftermath of maltreatment. Based on a literature review and findings of the previous follow-up study, we assume the following hypotheses:

* The HRQoL and mental health of children will be impaired following maltreatment even while controlling for others possible predictors of impaired HRQoL and mental health.
* We assume a dose-response relationship between severity of maltreatment and impaired HRQoL. Multiple maltreatment is hypothesized to have a larger impact then a single type of maltreatment.
* At baseline, HRQoL scores are hypothesized to be at a markedly low level. We assume a slight increase in HRQoL from baseline to first follow-up, but not a continuing increase to second follow-up.
* We assume differing trends for outcome variables in the aftermath of maltreatment and intend to analyze if types of trends are associated with clusters of risk and protective factors (cf. Chaffin, Bard, Hecht, & Silovsky, 2011).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* Outpatients
* Sexual abuse
* Physical maltreatment
* Psychological maltreatment
* Neglect
* Substantiated maltreatment
* Indicated maltreatment
* Aged 0-15 years at recruitment

Exclusion Criteria:

* telephone counseling
* Munchausen Syndrome by proxy
* Maltreatment not confirmed
* Aged 16 years and older at recruitment

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The sample is drawn from in- and outpatients reported to CPTs at University Children's Hospital Zurich and Children's Hospital Baden AG between July 2013 and August 2015.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Psychosocial development | Four years
  Normed and established instruments will be used for psychosocial assessment of children and caregivers. The assessment of child's development and well-being by primary caregivers will be complemented by child's self-assessment.
  Instruments:
  SON-R 2.5-7 (≥2.5 y.) DDST (0-5 years) KIDSCREEN-27 (≥8 y.) SDQ (11-17 y.) UCLA PTSD Index CDI (≥8 y.) CFT 1 (6-9.5 y.) or CFT 20-R (8.5-16 y.)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Jud, Dr., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital, Zurich, Canton of Zurich, Switzerland